CLINICAL TRIAL: NCT02629900
Title: The Effect of Time Restricted Feeding on Fat Mass in Overweight Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, PhD, University of Western Ontario, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 107401
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Weight Loss
Keywords: Weight Loss; Intermittent fasting
MeSH Terms: conditions — Weight Loss; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intermittent fasting group (Experimental): Participants will restrict their daily food intake (time restricted feeding) to an 8-hour time period between 1200 to 2000 hours. During the remaining 16-hour intermittent fasting period (2000 to 1200 hours) participants will be allowed to drink zero calorie beverages (diet soda pop, black coffee, tea, water, etc) in order to maintain normal hydration. There will be no attempt to restrict food intake. Rather simply to restrict the time period each day when food is consumed.
  Interventions: Behavioral: Time restricted feeding

INTERVENTIONS:
Behavioral: Time restricted feeding — Participants will consume their daily calories only between 12:00 and 20:00 for 4 weeks

SUMMARY:
Participants will complete a one-month intervention where they are will restrict their daily food intake to an 8-hour time period, i.e., between 1200 to 2000 hours. During the remaining 16-hour intermittent fasting period (2000 to 1200 hours) participants will be allowed to drink zero calorie beverages (diet soda pop, black coffee, tea, water, etc) in order to maintain normal hydration. There will be no attempt to restrict food intake. Rather simply to restrict the time period each day when food is consumed. Participants' body mass, fat mass, and non-fat mass will be monitored non-invasively using a weigh scale and densitometry via air displacement (Bod Pod) at 0, 2 and 4 weeks following the dietary intervention. Also, participants will be interviewed following the final body composition measure to assess whether or not they continued to follow the intermittent fasting approach.

DETAILED DESCRIPTION:
Participants (16 overweight women, BMI (Body mass index) ˃25, ages 18- 30 y)will complete a one-month intervention where they will restrict their daily food intake to an 8-hour time period, i.e., between 1200 to 2000 hours. During the remaining 16-hour intermittent fasting period (2000 to 1200 hours) participants will be allowed to drink zero calorie beverages (diet soda pop, black coffee, tea, water, etc) in order to maintain normal hydration. There will be no attempt to restrict food intake. Rather simply to restrict the time period each day when food is consumed. Participants' fat mass will be monitored non-invasively using densitometry (with a Bod Pod) prior to and following a 4 week intervention where the participants will eat their normal daily intake during an 8-hour period each day (1200 to 2000 hours). The Bod Pod measures body volume via air displacement and together with an accurate measure of body mass enables body density to be calculated (Density = mass/volume). Satisfaction, hunger, and fullness with the diet will be monitored on a weekly basis using a validated visual analog scale (Flit et al, 2000). Adherence to the diet will also be assessed on a weekly basis as the number of days the diet was followed. During the 16-hour fasting period participants will be able to drink as much of zero calorie beverages as they desire. On day 2, 7, 14, 21, & 28 participants will return to the lab at 8am (following a 12 hour fasting period) and both the acidity of their urine (using a urine dip stick) and their blood sugar (using a glucometer) will be tested. Following one month the participants will be allowed either to continue this eating pattern or revert to their prior 3 meal intake. After a month of self-regulation, the participants' fat mass will be measured again using the Bod Pod.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic participants between the ages of 18-30 years with body mass index ˃25 will be studied

Exclusion Criteria:

* Diabetic
* Pregnant
* Individuals with a history of fainting
* Low blood sugar
* Heart disease, migranes, or heart burn
* Participants less then 18 of age
* Anyone who for health or performance reasons should not skip breakfast will be excluded. These will be assessed by self report

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Fat mass change over 4 weeks period of intervention | 4 weeks
  Body fat mass change (%) will be measured using BodPod over the course of 4 weeks at 0, 2 and 4 weeks

SECONDARY OUTCOMES:
Non-fat mass change over 4 weeks period of intervention | 4 weeks
  Body non-fat mass (lean mass) (%) will be measured using BodPod over the course of 4 weeks at 0, 2 and 4 weeks
Urine acidity change over 4 weeks of intervention | 4 weeks
  Urine acidity will be measured following a 12 hours fasting at 0800 using a urine dip stick on days 2, 7, 14, 21, & 28
Blood sugar change over 4 weeks of intervention | 4 weeks
  Fasted blood sugar will be measured following a 12 hours fasting at 0800 using a finger prick glucometer (Free Style Lite) on days 2, 7, 14, 21, & 28
Diet satisfaction change over 4 weeks of intervention | 4 weeks
  Diet satisfaction will be monitored on a weekly basis using a validated visual analog scale (Flit et al, 2000)
Feeling of hunger change over 4 weeks of intervention | 4 weeks
  Hunger will be monitored on a weekly basis using a validated visual analog scale (Flit et al, 2000)
Feeling of fullness change over 4 weeks of intervention | 4 weeks
  Feeling of fullness will be monitored on a weekly basis using a validated visual analog scale (Flit et al, 2000)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lemon, PhD, Principal Investigator — Western University
Locations (1):
- Exercise Nutrition Research Laboratory, Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No